CLINICAL TRIAL: NCT02613754
Title: The Impact of Adding Contingency Management to Treatment as Usual for Disordered Gambling
Brief Title: Adding Contingency Management to Treatment as Usual for Disordered Gambling.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lethbridge (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Alberta Gambling Research Institute (Unknown)
Responsible Party: Principal Investigator, Darren R. Christensen, Chair in Gambling, Assistant Professor, University of Lethbridge
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSRC 2015-020
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Gambling, Pathological
MeSH Terms: conditions — Gambling | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management (Experimental): Contingency Management (CM+): This procedure is designed to reinforce treatment attendance, non-gambling behaviour, and study completion. Participants will earn points that will be recorded on vouchers that could be subsequently redeemed for gift cards at a variety of local businesses. Submission of evidence of gambling behaviour or non-attendance re-sets the point value for future vouchers to the starting level. This intervention is in addition to Treatment as Usual.
  Interventions: Behavioral: Contingency Management; Behavioral: Treatment as Usual
- Treatment as Usual (Active Comparator): Treatment as Usual (TAU): This is typically a semi-structured approach for delivering cognitive behavioural therapy addressing the participant's experiences, thoughts, and emotions relating to their gambling.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Contingency Management — See arm description.
  Arms: Contingency Management
Behavioral: Treatment as Usual — See arm description

SUMMARY:
The aim of this study is to conduct a trial to investigate the efficacy of adding Contingency Management (CM) to Treatment as Usual (TAU) for the treatment of Disordered Gambling. Results from this experiment will provide the first evidence of the additional efficacy of best-practice CM and whether it can be easily integrated into a clinical environment. Additionally, this study will correlate clinical outcomes with psychological measures and participant responses to develop new predictive treatment outcome measures.

DETAILED DESCRIPTION:
Hypothesis Behavioural approaches are direct and powerful ways of modifying problematic behaviours. The prediction is that adding best-practice CM treatments to TAU will reduce gambling behaviour and gambling urges to a greater degree than standard counselling practices.

Background Problematic gambling is a significant Canadian public health concern that causes harm to the gambler, their families, and society at large (Huang & Boyer, 2007). Approximately 4% of Albertans gamble in problematic ways resulting in significant financial losses, personal distress, relationship break-downs, and in some cases suicide (Williams et al., 2011; Problem Gambling Institute of Ontario, 2014). However, recent trends appear to show a decline in those seeking treatment despite the relatively consistent problem/disordered gambling prevalence rates (Williams et al., 2011). Further, 33% - 50% of treatment seekers drop out prior to the issue resolving (Leblonde et al., 2003), where those with the most severe gambling problems have the highest drop-out rates (ibid). One possible reason for these issues is the lack of immediate benefits clients gain from treatment attendance.

One treatment approach that provides immediate benefit for treatment attendance and superior treatment efficacy for substance and alcohol dependence is contingency management (Petry, 2010). Contingency management uses motivational incentives, typically vouchers that are exchangeable for retail goods and services, as rewards that participants receive for providing evidence of the target behavior and withholding them when the participant fails to perform the behaviour. This treatment has been used successfully in several countries in the treatment of various addictive substances (Garcia-Rodriguez et al., 2009; Peirce et al., 2006), and to promote healthy behaviours (Petry et al., 2011). Meta-analyses have consistently found contingency management to report improved clinical outcomes and the highest of treatment effect sizes (Dutra et al., 2010; Prendergast et al., 2006). Further, contingency management programs typically report a greater likelihood of program completion than standard care (Lott & Jencius, 2009), where the positive effects of the treatment persist many months after treatment completion (Petry & Martin, 2002).

Researchers are now suggesting that contingencies can be important mechanism in the treatment of gambling (Petry et al., 2006; Christensen, 2013), as the variable but regular nature of the receipt of gambling wins have been associated with the development of problematic gambling (Blaszczynski & Nower, 2002), where contingency management uses the same approach to reverse these associations. Moreover, recent research suggests that the development of non-gambling reinforcement can successfully compete with the gambling experience resulting in reductions in gambling behaviour and increases in alternative, and pro-social, behaviours (Jackson et al., 2013).

Although CM appears very successful, it has only been previously applied once to problematic gambling (West, 2008). However, there were issues with the pilot procedure (Christensen, 2013), as the program implemented was non-standard, notably the reinforcers were delayed, infrequent, of a low level, resulting in modest CM treatment outcomes (Petry, 2010). This proposal will use techniques that have been shown to improve the efficacy of a CM program. These are; 1) increasing the rate of incentives for sustained performance of the target behaviour and resetting following a lapse (Petry et al., 2006), 2) providing incentives at regular intervals (Christensen, 2013), 3) providing incentives as soon as practicable after evidence of the target behaviour is provided (Zeiler, 1977; Griffith et al., 2000), and 4) providing sufficiently meaningful incentives (Dallery et al., 2001). These additions to the standard CM procedure, which are typically used in successful treatments for substance dependence (Chopra et al., 2011), will hopefully improve the treatment efficacy of CM for disordered gamblers.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age, provide written consent, receive a diagnosis of disordered gambling, are primarily seeking treatment for disordered gambling, and speak English

Exclusion Criteria:

* Pharmacologically unmanaged psychiatric disorder that would impede counselling (e.g., psychosis), reports of neurological disorder(s), or injury resulting in a loss of consciousness greater than 10 minutes. Treatment as Usual participants will need to match CM+ participants on key measures (e.g., age, gender, education, gambling severity, substance use, psychiatric issues, comorbidities, treatment experience, ethnicity, and socio-economic status)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
The total number of sessions that a participant provided evidence of gambling abstinence in the study. | up to 12-weeks
  Gambling Abstinence

SECONDARY OUTCOMES:
The total number of sessions that a participant attended the study | up to 12-weeks
  Session Attendance
The total number of weeks that a participant attended the study. | up to 12-weeks
  Study Retention

CONTACTS AND LOCATIONS:
Overall Officials: Darren R Christensen, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- University of Lethbridge, Lethbridge, Alberta, Canada

REFERENCES:
- See also: Profile of Dr. Christensen — https://www.ulethbridge.ca/healthsciences/gambling-and-substance-use-studies